CLINICAL TRIAL: NCT02081976
Title: A Randomized, Controlled Trial to Study Effects of Periodontal Therapy in Primary Prevention of Cardiovascular Disease.
Brief Title: Periodontal Therapy in a Primary Prevention of Cardiovascular Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Macmillan Research Group UK (Industry)
Collaborators: Saibliss Healthcare Vision (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Mac/Saibliss 2120
Record Dates: First submitted 2014-03-06; First posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Periodontitis; Coronary Disease
MeSH Terms: conditions — Periodontitis; Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care Group (Active Comparator): Dental therapist providing standard periodontal treatment
  Interventions: Other: Standard Care Group
- Integrated Care Group (Experimental): a combined treatment approach of Dental Therapist, Dental Hygienist, Cardiologist along with counselor
  Interventions: Behavioral: Integrated Care Group

INTERVENTIONS:
Behavioral: Integrated Care Group — The group (TG) consisted of periodontal treatment comprising one session of supragingival scaling and personalized oral hygiene instructions, followed by one to four sessions of subgingival scaling and root planing (SRP) by quadrant, under local anesthesia, in a period of 14 days. Individuals were be followed monthly during the first 6 months. In the follow-up sessions, professional plaque removal, oral hygiene instructions, cardiac support along with counseling reinforcement were be provided.
  Arms: Integrated Care Group
Other: Standard Care Group — The group (TG) comprising one session of supragingival scaling followed by one to four sessions of subgingival scaling and root planing (SRP) by quadrant, under local anesthesia, in a period of 14 days.
  Arms: Standard Care Group

SUMMARY:
Cardiovascular diseases (CVD) are still considered the main cause of mortality and morbidity all over the world. In the last years, efforts have been made to define more effective therapeutic and preventive strategies.Periodontal diseases have been considered a probable risk factor for CVD with a great amount of evidence from observational studies. Although there are some interventional studies evaluating the systemic effects of periodontal therapy, there is little information regarding the impact of periodontal treatment on the prevention of cardiovascular events. To the best of our knowledge, there are no randomized controlled trials published to date assessing the effect of periodontal therapy in primary prevention of CVD.

ELIGIBILITY:
Inclusion Criteria:

* Individuals having at least 50% of their dentition with periodontal probing pocket depths N4 mm and
* With documented radiographic alveolar bone loss were included

Exclusion Criteria:

* Known systemic diseases
* History and/or presence of other infections
* Systemic antibiotic treatment in the preceding 3 months
* Treatment with any medication known to affect the serum level of inflammatory markers, lipids, or BP
* Pregnant or lactating females
* Allergy to tetracyclines

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Traditional cardiovascular risk markers (total cholesterol, LDL-C, HDL-C and triglycerides) | Change from baseline to six month

SECONDARY OUTCOMES:
High- and low-density lipoprotein cholesterol | Change from baseline to six month
cardiovascular risk scores (Framingham) | Change from baseline to six months

OTHER OUTCOMES:
Blood Pressure and Sugar | Change from baseline to six months

CONTACTS AND LOCATIONS:
Overall Officials: Neelam Maheshwari, BDS, Principal Investigator — Maheshwari Dental Clinic; Neha Sharma, PhD, Study Director — Macmillan Research Group
Locations (1):
- GyanSanjeevani, Jaipur, Rajasthan, India